CLINICAL TRIAL: NCT02414945
Title: Phase I/II Study Evaluating the Infusion of Tumor-Infiltrating Lymphocytes (TILs) & Low-Dose Interleukin-2 (IL-2) Therapy Following a Preparative Regimen of Non-myeloablative Lymphodepletion Using Cyclophosphamide & Fludarabine in Patients With Malignant Pleural Mesothelioma
Brief Title: TILs & Low-Dose IL-2 Therapy Following Cyclophosphamide and Fludarabine in Pleural Mesothelioma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILs-003-Meso
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tumor Infiltrating lymphocytes (TILs) (Experimental): Lymphodepleting preparative regimen: Cyclophosphamide, intravenously, at 60mg/kg/day x 2 days, and Fludarabine, intravenously at 25mg/m2/day x 5 days
  Autologous tumor infiltrating lymphocytes (TILs): Intravenously at 1x10^10 - 1.6x10^11 cells
  Low-dose interleukin-2: Subcutaneously at 125,000 IU/kg per day, for 2 weeks (2 days rest between each week).
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Autologous tumor infiltrating lymphocytes (TILs); Biological: Interleukin-2

INTERVENTIONS:
Drug: Cyclophosphamide
  Other Names: Procytox
Drug: Fludarabine
  Other Names: Fludara
Biological: Autologous tumor infiltrating lymphocytes (TILs)
Biological: Interleukin-2
  Other Names: Proleukin

SUMMARY:
This is a phase I and II clinical study for patients with malignant pleural mesothelioma (a type of cancer affecting the lining of the lung). Patients will receive an infusion (given by vein) of autologous tumor infiltrating lymphocytes (TILs). TILs are a type of white blood cells that recognizes tumor cells and enter them which causes the tumor cells to break down.

Prior to the cell infusion, patients will receive a two drugs cyclophosphamide and fludarabine to prepare the body to receive the TILs. After cell infusion, patients will receive low-dose interleukin-2 therapy. This study will see how safe and useful this regimen is in treating malignant pleural mesothelioma.

DETAILED DESCRIPTION:
The investigational infusion product consists of autologous, in vitro-expanded tumor-infiltrating lymphocytes (TILs). The target number of cells for infusion is between 1 x 1010 and 1.6 x 1011. The cells are given intravenously over a 20-30 minute infusion.

Prior to infusion of TILs, patients will receive a preparative regimen of cyclophosphamide (60 mg/kg/day x 2 days intravenously) and fludarabine (25 mg/m2/day x 5 days intravenously).

After the cell infusion, patients will receive low-dose interleukin-2 (IL-2) therapy (125,000 IU/kg/day subcutaneously for 2 weeks with a 2 day break between each week. The goal for the total number of doses is 9-10).

Because confusion is a possible side effect of IL-2 administration, a Durable Power of Attorney will be signed by the patient to identify a surrogate to make decisions if a patient becomes unable to make decisions.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign and date the informed consent form.
* Must have measurable stage I-IV malignant pleural mesothelioma at the time of investigational treatment.
* May have 3 or fewer asymptomatic brain metastases.
* Patient age: ≥ 18 years.
* Clinical performance status of ECOG 0 or 1.
* Life expectancy > 3 months from the date of consent.
* Laboratory analyses of tumor-infiltrating lymphocytes (TILs) from the patient must demonstrate that the TILs are suitable for use in protocol treatment
* More than 30 days has elapsed since any prior systemic therapy at the time of the cell infusion, or more than six weeks since prior nitrosurea therapy. All toxicities must have recovered to a grade 1 or less. Patients may have undergone minor surgical procedures with the past 3 weeks, as long as all toxicities have recovered to grade 1 or less
* Adequate organ function
* Women of child-bearing potential must have a negative pregnancy test. Patients of both genders must be willing to practice birth control during treatment and for 6 months post completion of IL-2 treatment.
* Patients must have adequate respiratory function in the opinion of the treating thoracic physician

Exclusion Criteria:

* Ongoing or prior use systemic steroid therapy within 4 weeks before the TILs infusion will be excluded.
* Known HIV positive patients will be excluded.
* Active hepatitis B or hepatitis C, syphilis, or HTLV will be excluded.
* Must not have any active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, uncontrolled psychiatric disorders, or other conditions that may affect compliance with the trial.
* Must have no active underlying cardiac illnesses defined by positive stress test, LVEF <40% or ongoing life threatening arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Total number of adverse events for each event reported and the severity and attribution to study therapy of each event | 5 years
  To determine the feasibility and safety of chemotherapy in combination with infusion of tumor-infiltrating lymphocytes followed by low-dose interleukin-2 in patients with malignant pleural mesothelioma.

SECONDARY OUTCOMES:
Percentage of patients with a clinical response to the study treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Butler, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada